CLINICAL TRIAL: NCT03380884
Title: Vibration Therapy as a Rehabilitation Intervention for Postural Training and Fall Prevention After Distal Radius Fracture in Elderly Patients: A Randomized Controlled Trial
Brief Title: Vibration Therapy as a Rehabilitation Intervention for Postural Training and Fall Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ronald Man Yeung WONG, Resident Doctor, Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017.447
Record Dates: First submitted 2017-11-30; First posted 2017-12-21 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Distal Radius Fracture; Fall Patients
Keywords: Distal Radius Fracture, Osteoporosis, Vibration Therapy
MeSH Terms: conditions — Wrist Fractures; Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group will remain in their habitual life style and no vibration used
- Vibration Group (Experimental): The intervention group will undergo Low-magnitude high-frequency vibration (LMHFV) at 35Hz, 0.3g (peak to peak magnitude), displacement of <0.1mm, 20 min/day, at least 3 times per week, for 6 months in community centres
  Interventions: Device: Low-magnitude high-frequency vibration (LMHFV)

INTERVENTIONS:
Device: Low-magnitude high-frequency vibration (LMHFV) — Low-magnitude high-frequency vibration (LMHFV) is a biophysical intervention that provides non-invasive, systemic mechanical stimulation and has been reported to have no adverse effect.
  Arms: Vibration Group

SUMMARY:
The occurrence of distal radius fractures is well known to be a sentinel event as these fractures are associated with 2 to 4 times increased risk of subsequent hip fractures in elderly patients. Studies have shown a significantly increased degree of postural sway in these patients, which is strongly associated with recurrent falls. The latest Cochrane systematic review also shows a lack of evidence on the effectiveness of current rehabilitation interventions.

Low-magnitude high-frequency vibration (LMHFV) is a biophysical intervention that provides non-invasive, systemic mechanical stimulation and has been shown to improve muscle strength and balancing abilities in healthy, independent and active elderly women in our previous clinical study. Our animal studies have also shown LMHFV promoting myogenic proliferation and hypertrophy, muscle contractibility, and increased fast-fiber switching to muscle fiber type IIA.Previous rehabilitation studies have used clinical functional performance tests, which lack sensitivity and specificity in predicting impaired postural control. The Biodex Balance System SD consists of a dynamic balance platform interfaced with computer software, which offers objective and reliable tests for postural stability and fall risk.

This study is a single-blinded, prospective randomized controlled trial to investigate the effect of 6 months of LMHFV after a distal radius fracture in elderly patients. Patients will be recruited and randomized to control or LMHFV group by envelope drawing of computer-generated random numbers. The intervention group will undergo LMHFV at 35Hz, 0.3g (peak to peak magnitude), displacement of <0.1mm, 20 min/day, at least 3 days/week for 6 months in community centres. Control group will remain in their habitual life style and no vibration used. Outcome assessments will be performed at baseline 0 days, 6 weeks, 3 months and 6 months. Outcome assessor and statistician will be blinded to group allocation.

The primary outcome is the effect of LMHFV on postural stability. The Biodex Balance System SD is used to measure the static and dynamic ability of the subjects to maintain the center of balance. Secondary outcomes are the occurrence of fall for the patients in both groups, the health-related quality of life (SF-36), and Timed Up and Go test for basic mobility skills.

DETAILED DESCRIPTION:
Distal Radius Fractures and Medico-socioeconomic Impact

Fractures of the distal radius account for approximately 380,000 fractures in the United States each year and occur in 15% of women older than 50 years of age. These fractures are a particular health concern amongst the elderly, who are at risk of fragility fractures, and are associated with long-term functional impairment, pain and a variety of complications. Over the past 10 years, there has been increased popularity of surgical interventions for the treatment of distal radius fractures, especially with the introduction of volar locking plates in 2000. Current medical costs for distal radius fractures are estimated to exceed USD 535 million each year and projected to rise as the incidence and use of internal fixation increases.

The Concept of Impaired Postural Stability and Prevention of Fall

The occurrence of distal radius fractures is well known to be a sentinel event as these fractures are associated with 2 to 4 times increased risk of subsequent hip fractures in elderly patients. This is an important concept as it is well established that these patients have an increased risk of falling. Fall prevention is therefore crucial to decrease further morbidity and mortality. Studies have shown a significantly increased degree of postural sway in patients with distal radius fractures, in both anteroposterior and lateral directions, which is strongly characterized in older subjects for recurrent falls. A recent study has also revealed that older adults have significantly impaired postural stability by using objective measurements from computerized instruments. Despite on-going studies on distal radius fractures, the latest Cochrane systematic review shows a lack of evidence on the effectiveness of current rehabilitation interventions. The American Academy of Orthopaedic Surgeons (AAOS) position statement also recommends patients with fragility fractures to undergo evaluation of osteoporosis and treatment to prevent future fractures. Notably, there are no recommendations on the role of balance training or physical conditioning. Consequently, the evaluation and treatment of fall risks have been largely overlooked. Further research that target rehabilitation and treat postural instability after distal radius fracture to reduce fall rates are therefore warranted.

Low-magnitude High-Frequency Vibration as a Rehabilitation Intervention to Improve Postural Instability and Prevent Fall

Low-magnitude high-frequency vibration (LMHFV) is a biophysical intervention that provides non-invasive, systemic mechanical stimulation and has been shown to improve muscle strength and balancing abilities in healthy, independent and active elderly women in our previous institute's study. Furthermore, our animal studies have also shown the ability of LMHFV to promote myogenic proliferation and hypertrophy, muscle contractibility, and increase fast-fiber switching to muscle fiber type IIA compared with control. Numerous other studies have reported whole body vibration to have positive effects on blood circulation in lower extremities and enhanced muscle performance including muscle strength in the elderly.

Previous rehabilitation studies have mainly used clinical functional performance tests, which lack sensitivity and specificity in predicting impaired postural control in osteoporotic patients. Therefore, the use of more objective measures to assess instability and fall risk derived from computerized instruments have been recommended. The Biodex Balance System SD (Biodex Medical Systems Inc, Shirley, NY) consists of a dynamic balance platform interfaced with computer software that provides up to 20° tilt from horizontal in a 360° range of motion. The system offers objective and reliable tests for postural stability and fall risk, which have been shown in multiple studies and in elderly patients.

In order to provide effective rehabilitation regimens for our patients, the validation of our interventions using objective outcomes is essential. To our knowledge, this is the first study to use an objective device to assess and validate our rehabilitation tool to prevent falls in patients after a distal radius fracture.

ELIGIBILITY:
Inclusion Criteria:

* 1) aged 60 or above
* 2) fracture distal radius after 6 weeks to 3 months
* 3) injury was due to unintentional fall.

Exclusion Criteria:

* 1) medical condition causing balance disturbance
* 2) participated in supervised regular exercise or physiotherapy for twice a week or more
* 3) Activities of Daily Living (ADL) dependent
* 4) malignancy
* 5) medications or condition that affect metabolism of the musculoskeletal system e.g. bisphosphonates

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Effect of LMHFV on postural stability | 0 days, 6 weeks, 3 months and 6 months. Change is being assessed
  To assess the postural stability, the Biodex Balance System SD is used to measure the ability of the subjects to maintain the center of balance. The Biodex Balance System SD has been shown to be a reliable tool for objective assessment of postural stability in several studies for elderly patients.

SECONDARY OUTCOMES:
Occurrence of fall for the patients in both groups | 0 days, 6 weeks, 3 months and 6 months. Change is being assessed
  To assess the occurrence of fall, subjects are required to self-report these events via a fall calendar, which has to be returned at every follow-up visit. Calendar reporting has been well proven to be reliable for fall studies
Health-related quality of life | 0 days, 6 weeks, 3 months and 6 months. Change is being assessed
  Health-related quality of life with a validated Chinese Version of the 36-Item Short-Form Health Survey (SF-36) will be used. All scores range from 0 to 100 with a higher score indicating better quality of life.
Timed Up and Go (TUG) test | 0 days, 6 weeks, 3 months and 6 months. Change is being assessed
  Timed Up and Go (TUG) test will be used to test the basic mobility skills.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Man Yeung Wong, Principal Investigator — Prince of Wales Hospital, Sha Tin, Hong Kong
Locations (1):
- Department of Orthopaedics and Traumatology, Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burge R, Dawson-Hughes B, Solomon DH, Wong JB, King A, Tosteson A. Incidence and economic burden of osteoporosis-related fractures in the United States, 2005-2025. J Bone Miner Res. 2007 Mar;22(3):465-75. doi: 10.1359/jbmr.061113. PMID 17144789
- [Background] Karantana A, Downing ND, Forward DP, Hatton M, Taylor AM, Scammell BE, Moran CG, Davis TR. Surgical treatment of distal radial fractures with a volar locking plate versus conventional percutaneous methods: a randomized controlled trial. J Bone Joint Surg Am. 2013 Oct 2;95(19):1737-44. doi: 10.2106/JBJS.L.00232. PMID 24088965
- [Background] Mellstrand-Navarro C, Pettersson HJ, Tornqvist H, Ponzer S. The operative treatment of fractures of the distal radius is increasing: results from a nationwide Swedish study. Bone Joint J. 2014 Jul;96-B(7):963-9. doi: 10.1302/0301-620X.96B7.33149. PMID 24986952
- [Background] Shauver MJ, Yin H, Banerjee M, Chung KC. Current and future national costs to medicare for the treatment of distal radius fracture in the elderly. J Hand Surg Am. 2011 Aug;36(8):1282-7. doi: 10.1016/j.jhsa.2011.05.017. Epub 2011 Jun 25. PMID 21705154
- [Background] Louer CR, Boone SL, Guthrie AK, Motley JR, Calfee RP, Wall LB. Postural Stability in Older Adults with a Distal Radial Fracture. J Bone Joint Surg Am. 2016 Jul 20;98(14):1176-82. doi: 10.2106/JBJS.15.00963. PMID 27440565
- [Background] Daruwalla ZJ, Huq SS, Wong KL, Nee PY, Leong KM, Pillay KR, Murphy DP. Hip fractures, preceding distal radius fractures and screening for osteoporosis: should we be screening earlier? A minimum 10-year retrospective cohort study at a single centre. Osteoporos Int. 2016 Jan;27(1):361-6. doi: 10.1007/s00198-015-3375-8. Epub 2015 Oct 28. PMID 26510846
- [Background] Kelsey JL, Prill MM, Keegan TH, Tanner HE, Bernstein AL, Quesenberry CP Jr, Sidney S. Reducing the risk for distal forearm fracture: preserve bone mass, slow down, and don't fall! Osteoporos Int. 2005 Jun;16(6):681-90. doi: 10.1007/s00198-004-1745-8. Epub 2004 Oct 26. PMID 15517189
- [Background] Crilly RG, Delaquerriere Richardson L, Roth JH, Vandervoort AA, Hayes KC, Mackenzie RA. Postural stability and Colles' fracture. Age Ageing. 1987 May;16(3):133-8. doi: 10.1093/ageing/16.3.133. PMID 3604793
- [Background] Handoll HH, Elliott J. Rehabilitation for distal radial fractures in adults. Cochrane Database Syst Rev. 2015 Sep 25;2015(9):CD003324. doi: 10.1002/14651858.CD003324.pub3. PMID 26403335
- [Background] Khazzani H, Allali F, Bennani L, Ichchou L, El Mansouri L, Abourazzak FE, Abouqal R, Hajjaj-Hassouni N. The relationship between physical performance measures, bone mineral density, falls, and the risk of peripheral fracture: a cross-sectional analysis. BMC Public Health. 2009 Aug 18;9:297. doi: 10.1186/1471-2458-9-297. PMID 19689795
- [Background] Leung KS, Li CY, Tse YK, Choy TK, Leung PC, Hung VW, Chan SY, Leung AH, Cheung WH. Effects of 18-month low-magnitude high-frequency vibration on fall rate and fracture risks in 710 community elderly--a cluster-randomized controlled trial. Osteoporos Int. 2014 Jun;25(6):1785-95. doi: 10.1007/s00198-014-2693-6. Epub 2014 Mar 28. PMID 24676848
- [Background] Cheung WH, Li CY, Zhu TY, Leung KS. Improvement in muscle performance after one-year cessation of low-magnitude high-frequency vibration in community elderly. J Musculoskelet Neuronal Interact. 2016 Mar;16(1):4-11. PMID 26944817
- [Background] Guo AY, Leung KS, Qin JH, Chow SK, Cheung WH. Effect of Low-Magnitude, High-Frequency Vibration Treatment on Retardation of Sarcopenia: Senescence-Accelerated Mouse-P8 Model. Rejuvenation Res. 2016 Aug;19(4):293-302. doi: 10.1089/rej.2015.1759. Epub 2016 Feb 19. PMID 26608404
- [Background] Sun KT, Leung KS, Siu PM, Qin L, Cheung WH. Differential effects of low-magnitude high-frequency vibration on reloading hind-limb soleus and gastrocnemius medialis muscles in 28-day tail-suspended rats. J Musculoskelet Neuronal Interact. 2015 Dec;15(4):316-24. PMID 26636277
- [Background] Cheung WH, Mok HW, Qin L, Sze PC, Lee KM, Leung KS. High-frequency whole-body vibration improves balancing ability in elderly women. Arch Phys Med Rehabil. 2007 Jul;88(7):852-7. doi: 10.1016/j.apmr.2007.03.028. PMID 17601464
- [Background] Roelants M, Verschueren SM, Delecluse C, Levin O, Stijnen V. Whole-body-vibration-induced increase in leg muscle activity during different squat exercises. J Strength Cond Res. 2006 Feb;20(1):124-9. doi: 10.1519/R-16674.1. PMID 16503671
- [Background] de Groot MH, van der Jagt-Willems HC, van Campen JP, Lems WF, Lamoth CJ. Testing postural control among various osteoporotic patient groups: a literature review. Geriatr Gerontol Int. 2012 Oct;12(4):573-85. doi: 10.1111/j.1447-0594.2012.00856.x. Epub 2012 Jun 4. PMID 22672622
- [Background] Broglio SP, Sosnoff JJ, Rosengren KS, McShane K. A comparison of balance performance: computerized dynamic posturography and a random motion platform. Arch Phys Med Rehabil. 2009 Jan;90(1):145-50. doi: 10.1016/j.apmr.2008.06.025. PMID 19154841
- [Background] Arifin N, Abu Osman NA, Wan Abas WA. Intrarater test-retest reliability of static and dynamic stability indexes measurement using the Biodex Stability System during unilateral stance. J Appl Biomech. 2014 Apr;30(2):300-4. doi: 10.1123/jab.2013-0130. Epub 2013 Jul 20. PMID 23878204
- [Derived] Wong RMY, Ho WT, Tang N, Tso CY, Ng WKR, Chow SK, Cheung WH. A study protocol for a randomized controlled trial evaluating vibration therapy as an intervention for postural training and fall prevention after distal radius fracture in elderly patients. Trials. 2020 Jan 16;21(1):95. doi: 10.1186/s13063-019-4013-0. PMID 31948477

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT03380884/Prot_SAP_000.pdf